CLINICAL TRIAL: NCT04190225
Title: Individually Tailored Physical Activity Intervention for Latina Adolescents: Chicas Fuertes
Brief Title: Physical Activity Intervention for Adolescent Girls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Brown University (Other)
Responsible Party: Principal Investigator, Britta Larsen, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 182070; R01NR017876 (NIH)
Record Dates: First submitted 2019-11-20; First posted 2019-12-09 (Actual); Results first posted 2025-05-04 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Physical Activity
Keywords: physical activity; adolescents; teenagers; Latina
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: 1:1 treatment: control
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-technology physical activity intervention (Experimental): Digital/social media
  Interventions: Behavioral: Digital/social media intervention
- Control (No Intervention): Control group receives a Fitbit but none of the intervention components.

INTERVENTIONS:
Behavioral: Digital/social media intervention — Participants will receive individual counseling, access to an individually tailored website, guided goal setting via texts, access to a study Instagram account, and a wearable tracker (Fitbit)
  Arms: Multi-technology physical activity intervention

SUMMARY:
This study will conduct a randomized trial to evaluate the efficacy of a theory-based, individually tailored, multi-technology intervention on increasing physical activity in Latina adolescents, compared to a control group receiving only a physical activity tracker (a Fitbit). The investigators will recruit adolescent (age 13-18) Latinas (N=200) who are currently underactive to participate in the 12-month trial. Those randomized to the Intervention arm will receive a one-on-one counseling session and access to an individually tailored multi-media website. Key intervention components will be reinforced through text messaging to aid goal setting, a physical activity tracker (Fitbit) to set goals, track and log activity, and access to a study Instagram account to reinforce exposure to web content. The primary outcome will be increases in moderate-to-vigorous activity between baseline and 6 months. Secondary outcomes will include changes in activity at 12 months, potential mediators of the intervention, costs of delivering the intervention, behavior change trajectories from continuous data from Fitbits, potential moderators, and changes in physiological and psychological variables.

DETAILED DESCRIPTION:
Latina adolescents report low levels of physical activity, with only 3% meeting national physical activity guidelines, and are at high lifetime risk for conditions related to inactivity, such as obesity, metabolic syndrome, and diabetes. Interventions grounded in sound psychosocial theory and leveraging growing technology use in Latina adolescents are needed to reverse patterns of inactivity, establish healthy lifetime habits and reduce widening disparities. The research team has developed and tested individually tailored, culturally adapted web-based interventions to increase moderate-to-vigorous physical activity (MVPA) for Latinos, which significantly increased MVPA in adult Latino men and women. In a recent pilot study (R03NR014329), this intervention was adapted based on formative interviews to make it appropriate for Latina adolescents and tested it in a single-arm pilot trial (N=21). After 12 weeks, retention was high (90.5%) and self-reported MVPA increased from 24.7(26.11) minutes/week at baseline to 79.4(46.8) at follow up (p<0.001), suggesting good potential efficacy. In closeout interviews, girls expressed a preference to increase audiovideo components of the website and to incorporate other mobile-health technologies, such as texting, smartphone apps, social media, and wearables. Thus, the aim of this study is to conduct a randomized controlled trial (N=200) of an individually tailored, theory-based, multi-technology intervention to increase MVPA in Latina adolescents. The intervention will comprise a counseling session to teach behavior change techniques, an interactive multimedia website with individually tailored content based on principles of the Transtheoretical Model and Social Cognitive Theory, a wearable tracker and smartphone app to reinforce key behavior change techniques, connection with a study Instagram account to reinforce exposure to intervention content, and automated text messages guide continued goal setting. Participants will be randomly assigned to receive the intervention or only a wearable tracker with smartphone app. Activity will be measured at baseline and six-month follow-up using well-established MVPA measures (accelerometers and the 7-Day Physical Activity Recall Interview). It is hypothesized that those randomized to receive the intervention will show significantly greater increases in MVPA at six months than those in the control group. The investigators will also evaluate whether changes in MVPA are mediated by changes in targeted psychosocial constructs (e.g. self-efficacy, social support) or engagement with technology, assess longer-term changes in MVPA at 12 months, and evaluate whether intervention effects are moderated by baseline personal and environmental variables (e.g. age, BMI, neighborhood environment). Costs to deliver the intervention (e.g. staff time, materials, overhead) will be tracked to evaluate costs and cost-effectiveness of both study arms, and the investigators will track contact time to assess whether staff contact is related to study outcomes. The investigators will also explore trajectories of daily activity in both the intervention and control groups using continuous data from wearable trackers. The proposed study will promote a critical preventive health behavior, physical activity, in Latina adolescents using technologies that are pervasive in this high risk, quickly growing population and highly scalable, laying the groundwork for cost-effective, broad reaching interventions with great potential for preventing chronic disease and promoting health and wellbeing throughout the lifespan.

ELIGIBILITY:
Inclusion Criteria:

* self identify as Latina
* 13-18 years old
* read, write, speak English
* under active (participating in <150 minutes of moderate to vigorous physical activity per week)
* regular access to the Internet (at least 2 times per week)
* regular access to a cell phone that can send and receive text messages

Exclusion Criteria:

* inability to safely engage in physical activity, as determined by the Physical Activity Readiness Questionnaire
* BMI > 45
* Plan to move from the area within 12 months

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 160 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2024-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Britta Larsen, PhD, Principal Investigator — UCSD
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Larsen B, Greenstadt E, Olesen B, Osuna L, Godino J, Marcus B, Dunsiger S, Meyer D, Zive M. A multiple technology-based physical activity intervention for Latina adolescents in the USA: randomized controlled trial study protocol for Chicas Fuertes. Trials. 2022 Feb 23;23(1):176. doi: 10.1186/s13063-022-06105-2. PMID 35197106

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 306 individuals were screened for eligibility. Of these 188 were eligible. Primary reasons for ineligibility were being too active (65), being outside the age range (24), BMI too high (4), not having access to technology (2), not living in the area (4), not speaking English (3), not being female or Latina (5), and other (10). Of the 188 eligible, 28 declined to participate after learning more about the study.
Period: Overall Study
Arm/Group | Multi-technology Physical Activity Intervention | Control
Started | 77 | 83
Completed | 70 | 78
Not Completed | 7 | 5
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Unrelated health condition | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Multi-technology Physical Activity Intervention | Control | Total
Number analyzed (Participants) | 77 | 83 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.8 (1.7) | 15.9 (1.5) | 15.9 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 83 | 160
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 77 | 83 | 160
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 35 | 33 | 68
  More than one race | 8 | 4 | 12
  Unknown or Not Reported | 31 | 43 | 74
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.2 (5.5) | 25.2 (6.6) | 25.7 (6.1)
Primary Language [Count of Participants; unit: Participants]
  Mostly Spanish | 4 | 6 | 10
  Spanish and English equally | 21 | 31 | 52
  English more than Spanish | 47 | 37 | 84
  Only English | 5 | 9 | 14
Generation Status [Count of Participants; unit: Participants]
  First | 6 | 7 | 13
  Second | 53 | 57 | 110
  Third | 18 | 19 | 37
Parent Education [Count of Participants; unit: Participants]
  High school or less | 42 | 44 | 86
  At least some college | 35 | 39 | 74
Family Income [Count of Participants; unit: Participants]
  <$50,000 | 45 | 54 | 99
  ≥$50,000 | 32 | 29 | 61
Number of children in home [Mean (Standard Deviation); unit: number of children] | 2.01 (1.2) | 1.93 (1.2) | 1.97 (1.2)
Neighborhood Walkability - Street Connectivity [Mean (Standard Deviation); unit: units on a scale] — The Street Connectivity sub-scale of the Neighborhood Environment Walkability Scale for Youth (NEWS-Y) has 3 items rated 1-4 (agree/disagree). Scores are averaged, with higher scores indicating higher perceived street connectivity.
  units on a scale | 2.83 (0.6) | 2.84 (0.6) | 2.83 (0.6)
Neighborhood Environment [Mean (Standard Deviation); unit: units on a scale] — The Physical Activity Neighborhood Environment scale (PANES) is an 8-item measure used to measure neighborhood walkability. Scoring ranges from 0-6, with higher numbers indicating higher walkability.
  units on a scale | 4.96 (1.2) | 4.57 (1.4) | 4.77 (1.3)
Physical Activity Enjoyment [Mean (Standard Deviation); unit: units on a scale] — The Physical Activity Enjoyment Scale (PACES) consists of 18 items rated on a 7-point Likert scale, and it measures enjoyment of physical activity. The total scoring range is 18-126. Results reported are an average score across the 18 items (1-7 range), with higher scores indicating greater enjoyment.
  units on a scale | 4.67 (0.92) | 5.03 (0.93) | 4.86 (0.94)
Depressive Symptoms [Mean (Standard Deviation); unit: units on a scale] — Depressive Symptoms were measured using the Center for Epidemiologic Studies Depression Scale (CES-D-10), a 10-item scale with response options ranging from "rarely or none of the time" (0) to "all of the time" (3). Total scores can range from 0 to 30, with a higher score indicating greater presence of depressive symptoms.
  units on a scale | 10.62 (3.9) | 11.14 (4.7) | 10.9 (4.3)
Self-Efficacy for Physical Activity [Mean (Standard Deviation); unit: units on a scale] — This 5-item instrument measures self efficacy to exercise when facing various barriers to exercise. There are 4 response options ranging from "Not at all confident" to "Very confident." Total scoring range is from 5-20, with an average taken across the 5 items resulting in an average score of 1-4. Higher numbers indicate higher self efficacy.
  units on a scale | 1.98 (0.54) | 2.03 (0.46) | 2.01 (0.50)
Social Support for Exercise [Mean (Standard Deviation); unit: units on a scale] — The Social Support for Exercise scale (SSE) is frequently used among Hispanic populations. The 13-item survey is comprised of statements, which participants rate on a 1-5 Likert scale, with a scoring range from 13-65. A higher score indicates higher levels of social support for exercise.
  units on a scale | 20.5 (13.4) | 24.2 (16.7) | 22.4 (15.3)
Maternal Support for Exercise [Mean (Standard Deviation); unit: units on a scale] — The 26-item Maternal Support for Exercise questionnaire is administered to Latina mother-daughter dyads. The mothers' version rates how often they engaged in behaviors supporting their daughters' physical activity, and the daughters' version rates how often their mothers' engaged in these aforementioned behaviors. Each of the 26 items is rated using a 5-point Likert response option ranging from 1 = never to 5 = always/daily. Associations between mother and daughter dyads' scores are calculated, with higher scores indicating higher maternal support.
  units on a scale | 2.46 (0.75) | 2.55 (0.64) | 2.51 (0.69)
Exercise Stage of Change [Count of Participants; unit: Participants]
  Pre-contemplation | 3 | 1 | 4
  Contemplation | 10 | 12 | 22
  Preparation | 64 | 70 | 134
ActiGraph Physical Activity [Median (Inter-Quartile Range); unit: minutes of activity] | 0 [0 to 24] | 0 [0 to 26] | 0 [0 to 24]
Self-Reported Physical Activity [Median (Inter-Quartile Range); unit: minutes of activity] | 119 [62.5 to 185] | 120 [48.8 to 235] | 120 [55 to 205]
Daily Steps [Mean (Standard Deviation); unit: average daily steps across one week] | 5196 (3116) | 5275 (3191) | 5222 (3359)
Land-use mix - NEWS-Y [Mean (Standard Deviation); unit: units on a scale] — The Land Use Mix sub-scale of the Neighborhood Environment Walkability Scale for Youth (NEWS-Y) has 20 items listing businesses in the neighborhood, each of which is rated for walking distance (1 = 5 minutes, 5 = 30+ minutes). Scores are reverse coded and averaged, with higher scores indicating higher walkability.
  units on a scale | 2.47 (0.62) | 2.37 (0.81) | 2.42 (0.73)
Recreation Facilities - NEWS-Y [Mean (Standard Deviation); unit: units on a scale] — the recreation facilities sub-scale of the Neighborhood Environment Walkability Scale for Youth (NEWS-Y) includes 14 recreation facilities which are rated 1-5 for walking proximity (1 = 5 minutes, 5 = 30+ minutes). Scores are reverse coded and averaged, with higher scores indicating higher walkability.
  units on a scale | 2.27 (0.68) | 2.21 (0.76) | 2.24 (0.72)
Residential Density - NEWS-Y [Mean (Standard Deviation); unit: units on a scale] — The Residential Density sub-scale of the Neighborhood Environment Walkability Scale for Youth (NEWS-Y) has 4 items describing types of housing, which are rated 1-5 for perceived commonness in their neighborhood (1 = none, 5 = all). Scores are weighted and summed, with totals ranging from 40 to 200. Higher scores indicate higher walkability.
  units on a scale | 112 (39.1) | 109 (40.3) | 111 (39.6)
Land use access - NEWS-Y [Mean (Standard Deviation); unit: units on a scale] — The land use access sub-scale of the Neighborhood Environment Walkability Scale for Youth (NEWS-Y) has 6 items describing walkability in the participant's neighborhood, which are rated from 1 (disagree) to 4 (agree). Scores are averaged, with higher scores indicating higher walkability.
  units on a scale | 2.94 (0.50) | 3.01 (0.50) | 2.98 (0.50)
Walking/cycling facilities - NEWS-Y [Mean (Standard Deviation); unit: units on a scale] — The walking/cycling facilities sub-scale of the Neighborhood Environment Walkability Scale for Youth (NEWS-Y) has 3 items describing facilities to walk or bike within the participant's neighborhood. Items are rated from 1 (disagree) to 4 (agree). Scores are averaged, with higher scores indicating greater walkability.
  units on a scale | 3.07 (0.59) | 3.05 (0.66) | 3.06 (0.63)
Neighborhood aesthetics - NEWS-Y [Mean (Standard Deviation); unit: units on a scale] — The neighborhood aesthetics sub-scale of the Neighborhood Environment Walkability Scale for Youth (NEWS-Y) has 4 items describing aesthetic elements of the participant's neighborhood. Items are rated from 1 (disagree) to 4(agree). Scores are averaged, with higher scores indicating better aesthetics and higher walkability.
  units on a scale | 2.74 (0.66) | 2.89 (0.73) | 2.82 (0.7)
Safety from traffic - NEWS-Y [Mean (Standard Deviation); unit: units on a scale] — The safety from traffic sub-scale of the Neighborhood Environment Walkability Scale for Youth (NEWS-Y) has 7 items describing pedestrian and automobile traffic safety in the participant's neighborhood. Items are rated from 1 (disagree) to 4 (agree). Scores are averaged, with higher scores indicating lower safety and lower walkability.
  units on a scale | 2.78 (0.45) | 2.79 (0.45) | 2.78 (0.45)
Safety from crime [Mean (Standard Deviation); unit: units on a scale] — The safety from crime sub-scale of the Neighborhood Environment Walkability Scale for Youth (NEWS-Y) has 6 items describing crime in the participant's neighborhood. Items are rated from 1 (disagree) to 4 (agree). Scores are averaged, with higher scores indicating higher crime and lower walkability.
  units on a scale | 2.26 (0.78) | 2.19 (0.75) | 2.22 (0.76)

OUTCOME MEASURES:

1. Primary Outcome: Objectively Measured Weekly Minutes of Activity
Description: The ActiGraph GT3X+ accelerometer will be the primary measure to assess objective changes in physical activity from baseline to 6 months. (waking hours only) to measure movement and intensity of activity
Time Frame: Baseline, 6 Months (MO)
Measure: Median (Inter-Quartile Range); unit: weekly minutes of activity
Arm/Group | Multi-technology Physical Activity Intervention | Control
Number analyzed (Participants) | 70 | 78
weekly minutes of activity | 64 [19 to 72] | 41 [7 to 76]
Statistical Analysis 1: Comparison: Multi-technology Physical Activity Intervention vs Control; Test type: Superiority; p = 0.04, quantile regression; Median Difference (Final Values) = 18.4, 95% CI 2-sided [4.67 to 37.28] — Median difference is not the difference in the two medians, but is the median of differences between groups (why it is 18.4 and not 23)

2. Primary Outcome: Self-Reported Weekly Minutes of Activity
Description: The 7-Day Physical Activity Recall (PAR) will also assess self-reported changes in physical activity from baseline to 6 months. The 7-Day PAR is an interviewer administered instrument that uses multiple strategies for increasing accuracy of participant recall regarding many types of activities such as time spent sleeping and moderate, hard, and very hard intensity activities. The 7-Day PAR is used across many studies assessing physical activity and has consistently demonstrated acceptable reliability, internal consistency, and congruent validity with other objective measures of activity levels.
Time Frame: Baseline, 6 Months (MO)
Measure: Median (Inter-Quartile Range); unit: minutes of activity per week
Arm/Group | Multi-technology Physical Activity Intervention | Control
Number analyzed (Participants) | 70 | 78
minutes of activity per week | 147 [96 to 181] | 124 [100 to 169]
Statistical Analysis 1: Comparison: Multi-technology Physical Activity Intervention vs Control; Test type: Superiority; p = 0.03, quantile regression; Median Difference (Final Values) = 23.5, 95% CI 2-sided [8.35 to 32.76]

3. Secondary Outcome: Objectively Measured Weekly Minutes Minutes of Activity
Description: weekly minutes of moderate-to-vigorous physical activity measured by ActiGraph accelerometer
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: weekly minutes of activity
Arm/Group | Multi-technology Physical Activity Intervention | Control
Number analyzed (Participants) | 65 | 70
weekly minutes of activity | 74 [32 to 120] | 37 [12 to 91]
Statistical Analysis 1: Comparison: Multi-technology Physical Activity Intervention vs Control; Test type: Superiority; p < .001, quantile regression

ADVERSE EVENTS:
Time Frame: 6 months
Description: Participants were asked to alert the study team of any injuries or adverse events experienced during the trial within 24 hours of experiencing them
Arm/Group | Multi-technology Physical Activity Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/83
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/83
Other Adverse Events (participants affected / at risk) | 0/77 | 0/83

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-04): https://cdn.clinicaltrials.gov/large-docs/25/NCT04190225/Prot_SAP_001.pdf
  • Informed Consent Form (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/25/NCT04190225/ICF_000.pdf